CLINICAL TRIAL: NCT06272721
Title: Investigation of the Association Between Hypothyroidism in Pregnancy and Neuropsychological Development in Children
Brief Title: Hypothyroidism in Pregnancy and Neuropsychological Development in Children
Acronym: OHPLDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6272
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Dysfunction; Pregnancy Related; Language Development

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Children of women with overt hypothyroidism during pregnancy (Other): 31 children undergoing neuropsychological testing for clinical practice, having their 31 mothers exhibited overt hypothyroidism during pregnancy.
  Interventions: Diagnostic Test: Griffiths Scale
- Group 2: Children of women without overt hypothyroidism during pregnancy (Active Comparator): 21 children undergoing neuropsychological testing outside of clinical practice, as their 21 mothers did not exhibit overt hypothyroidism during pregnancy.
  Interventions: Diagnostic Test: Griffiths Scale

INTERVENTIONS:
Diagnostic Test: Griffiths Scale — The Griffiths Mental Development Scales II are key tools for assessing children's psychomotor development from ages 0 to 6, praised for their strong psychometric properties. They evaluate various functional areas through six subscales, combining parental reports and direct observations of the child's behavior. The areas include locomotion, personal-social interaction, learning and language, eye-hand coordination, and performance, excluding the optional practical reasoning section for older children in this study. The Development Quotient (DQ), calculated by comparing mental and chronological ages, indicates developmental progress or delay, with an average score around 100 ± 15.

SUMMARY:
Thyroid dysfunction, particularly hypothyroidism and thyroid autoimmunity, impacts a significant proportion of pregnant women, affecting 3% and 17% respectively. The management of thyroid-stimulating hormone (TSH) levels is crucial, with subclinical hypothyroidism often defined by a TSH upper reference limit of 4 mU/L, and overt hypothyroidism by TSH levels above 10 mU/L and potentially low free thyroxine (FT4) levels. Levothyroxine (LT4) treatment is strongly advised for TSH levels above 10 mU/L, with the timing of intervention being critical during the first trimester for optimal fetal brain development.

Research shows that untreated maternal hypothyroidism can significantly impact the neuropsychological development of the child, affecting cognitive, verbal, and motor skills. Even subclinical maternal hypothyroidism has been associated with lower IQ and motor scores in children. Early pregnancy intervention is key, as treatment after the first trimester may not improve children's neurocognitive outcomes.

Regarding sensory and linguistic development, evidence is mixed, but recent studies suggest that maternal hypothyroidism can lead to expressive language delays. The Development Quotient (DQ) is used to assess cognitive and motor development in children, with the Griffiths Mental Development Scales II being a common tool.

This study aims to explore the effects of treated maternal hypothyroidism during pregnancy on children's neurodevelopment, focusing on learning and language. It includes 31 women diagnosed with hypothyroidism and a control group of 21 euthyroid women, along with their children. The study emphasizes the importance of early detection and treatment of maternal hypothyroidism for preventing adverse neurodevelopmental outcomes in offspring. Statistical analysis will be conducted using SPSS, with a focus on maternal-fetal outcomes and cognitive-neuropsychological outcomes, highlighting the significance of early intervention.

DETAILED DESCRIPTION:
Thyroid dysfunction is a not uncommon endocrine disorder during pregnancy, with hypothyroidism and thyroid autoimmunity affecting respectively 3% and 17% of expectant mothers. The value of thyroid-stimulating hormone (TSH) during pregnancy should be assessed in reference to a specific population and a trimester range, ideally defined by the reference laboratory or obtained from a similar population. When this is not possible, an upper reference limit of 4 mU/L (4 µIU/mL) may be used to define subclinical hypothyroidism. Elevated TSH values (above 10 mU/L (10 µIU/mL)) possibly associated with low levels of free thyroxine (FT4) define overt hypothyroidism. Current guidelines strongly recommend levothyroxine (LT4) therapy in women with TSH above 10 mU/L (10 µIU/mL), while recommendations regarding subclinical hypothyroidism are more debated and depend on antibody positivity. Regarding the timing of LT4 intervention, the most critical phase is the first trimester, as the fetal thyroid is fully functional after week 12, when thyroid organogenesis is complete. The consistent intake of thyroid hormones is crucial for brain maturation, influencing numerous aspects including migration, differentiation, and neural cell signaling. Data regarding the association between overt hypothyroidism and adverse pregnancy complications are quite solid. Gestational hypothyroidism has been linked to an increased risk of preterm birth, intrauterine growth restriction (IUGR) of fetuses, spontaneous abortion, and risk of fetal death, particularly when hypothyroidism was untreated or inadequately managed. Studies on the influence of maternal prenatal thyroid dysfunction show that it can alter cognitive, verbal, and motor abilities in children. Already in 1999, it was highlighted that children born to mothers with untreated hypothyroidism had a lower intelligence quotient (IQ). These negative effects have also been observed in subclinical hypothyroidism. Children of mothers with elevated TSH levels show reductions in intelligence and motor scores. Furthermore, lower intellectual development seems correlated with maternal TSH level, regardless of the presence of antibodies. Studies have also revealed that treatment of maternal hypothyroidism after the first trimester of pregnancy does not necessarily improve the neurocognitive abilities of children. This suggests that interventions are more effective if they occur in the early stages of pregnancy. Regarding sensory and linguistic development, the evidence is conflicting. Some studies have found no significant correlations, while others have observed that maternal hypothyroidism may be associated with delays in expressive language. A recent study showed a decrease in language scale scores in children born to mothers with overt hypothyroidism. This indicates that the balance of thyroid hormones during pregnancy is crucial for the optimal neurocognitive development of the child. The Development Quotient (DQ) is an index that measures cognitive and motor development in children, similar to the Intelligence Quotient (IQ), but specific for preschool and infant age. It includes tests that assess linguistic, motor, social, and problem-solving skills. A high score indicates normal or advanced development, while a low one may signal delays or the need for specific interventions. Among the tools to assess DQ, the Griffiths Mental Development Scales II are widely used for children from 0 to 6 years. These scales have six subscales that evaluate different functional areas, based on parent information and direct observations. The areas are: locomotion, personal-social interaction, learning and language, eye-hand coordination, performance, and practical reasoning (the latter not always assessed). The DQ is calculated by comparing the mental age with the chronological age of the child and is expressed as DQ. An average DQ stands at about 100 ± 15. The study will pay particular attention to specific neurocognitive areas such as learning and language. Furthermore, we will analyze the pregnancy outcome and complications in mothers. The aim of this study is to explore the connection between maternal hypothyroidism treated during pregnancy and the neurological development of the offspring, focusing on learning and language and examining related maternal obstetric complications. The study will include 31 women who were diagnosed with hypothyroidism and a control group of 21 euthyroid women. 31 children of hypothyroid women and 21 children of euthyroid women. The inclusion criteria encompass all women who were diagnosed with hypothyroidism - whether post-surgical or autoimmune, preexisting or newly diagnosed - presenting TSH values equal to or higher than 10 mU/L (10 µIU/mL) (n.v. 0.5-2.5) during pregnancy. The exclusion criteria applied to both groups involve the presence of uncontrolled liver, kidney, diabetic, neurological, and psychiatric comorbidities before conception, twin pregnancies, a history of alcohol consumption or smoking during pregnancy, and a history of infertility or assisted conception. The statistical analysis foresees that continuous data will be represented as mean ± standard deviation (SD), while categorical variables will be presented as frequency and percentage. In comparing baseline characteristics between groups, the Chi-square test will be used for categorical variables, while the independent Student's t-test will be applied for normally distributed continuous quantitative variables. The analysis of outcomes will be bifurcated into maternal-fetal outcomes and cognitive-neuropsychological outcomes. For comparisons between groups regarding outcomes, the Chi-square test will be used for categorical variables, the independent Student's t-test for normally distributed continuous quantitative variables, and the Mann-Whitney U test for non-normally distributed quantitative variables. A p-value of less than 0.05 will be considered statistically significant. Furthermore, a correlation analysis between two non-normally distributed quantitative variables will be conducted, where a p-value of less than 0.01 will be considered statistically significant. All statistical analyses will be performed using SPSS software (IBM) version 25

ELIGIBILITY:
Inclusion Criteria Group 1:

Women aged above 18 and not beyond 50; Diagnosed with hypothyroidism during pregnancy; TSH values equal to or greater than 10 mU/L during pregnancy; Children aged between 2 and 6 years born to mothers with overt hypothyroidism during pregnancy; Signature of consent.

Exclusion Criteria Group 1:

Presence of uncontrolled liver, kidney, diabetic, neurological, and psychiatric comorbidities prior to conception; Twin pregnancies; History of alcohol or smoking during pregnancy; History of infertility or assisted conception.

Inclusion Criteria Group 2:

Women aged above 18 and not beyond 50; Absence of hypothyroidism during pregnancy; Children aged between 2 and 6 years born to mothers without overt hypothyroidism during pregnancy; Signature of consent.

Exclusion Criteria Group 2:

Presence of uncontrolled liver, kidney, diabetic, neurological, and psychiatric comorbidities prior to conception; Twin pregnancies; History of alcohol or smoking during pregnancy; History of infertility or assisted conception.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-02-19 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
total development quotient measured using the Griffiths scale | 30 minuts
  Difference in the total Development Quotient (DQ) measured using the Griffiths scale, which evaluates different areas of neurodevelopment, between children born to mothers with overt hypothyroidism (TSH > 10 mIU/L) and children born to women without overt hypothyroidism.
  Difference in the total Development Quotient (DQ) measured using the Griffiths scale, which evaluates different areas of neurodevelopment, between children born to mothers with overt hypothyroidism (TSH > 10 mIU/L) and children born to women without overt hypothyroidism.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Pontecorvi, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy